CLINICAL TRIAL: NCT04856774
Title: A Multicenter, Open-Label, Phase Ib/II Trial of SHR-1701 Plus BP102 in Subjects With Selected Solid Tumors
Brief Title: Trial of SHR-1701 Plus BP102 in Subjects With Selected Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-II-207
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR -1701 + BP102 (Experimental)
  Interventions: Drug: SHR-1701；BP102

INTERVENTIONS:
Drug: SHR-1701；BP102 — Drug: SHR-1701 IV infusion
  Drug: BP102 IV infusion
  Phase Ib: SHR-1701 30mg/kg + BP102 15mg/kg Q3w as starting dose, until recommended phase 2 dose is determined.

SUMMARY:
The main purpose of this study was to assess the safety, tolerability, and efficacy when combining SHR-1701 and BP102 in participants with certain cancers. This study was conducted in 2 phases, Phase Ib and Phase II.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid malignancy that is metastatic or unresectable for which standard curative or palliative measures do not exist or are no longer effective (phase Ib)
2. Histologically or cytologically confirmed metastatic or locally advanced solid tumors of the selected indications. (Phase II).
3. .Life expectancy exceeds 12 weeeks;
4. The Eastern Cancer Cooperative Group (ECOG) has a performance score of 0 or 1;
5. Normal organ and marrow function;

Exclusion Criteria:

1. Has known active central nervous system (CNS) metastases. Subjects with previously treated brain metastases may participate provided they are stable.
2. A history of human immunodeficiency virus (HIV) infection is known, or has an active autoimmune disease.
3. History of interstitial lung disease or pneumonia requiring oral or intravenous steroids.
4. Has moderate or severe cardiovascular disease;
5. Active HBV(hepatitis B) or HCV (Hepatitis C virus)-infected subjects;
6. Any other malignancies within 5 years except for those with negligible risk of metastasis or death.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
recommended phase 2 dose (Phase Ib) | At the end of Cycle 2 (each cycle is 21 days)
Objective response rate (ORR) | 2 years

SECONDARY OUTCOMES:
Dose Limiting Toxicity (DLT) (Phase 1b) | At the end of Cycle 2 (each cycle is 21 days)
Number of participants with treatment emergent adverse events (TEAEs) | For each participant, from the first dose till 90 days after the last dose
Number of participants with treatment emergent serious adverse events (SAEs) | For each participant, from the first dose till 90 days after the last dose
ORR | 2 years
Duration of response (DOR) | 2 years
Disease control rate (DCR) | 2 years
Time to response(TTR) | 2 years
Progression-free survival (PFS) | 2 years
Overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangzhou, China